CLINICAL TRIAL: NCT00819910
Title: Rosiglitazone And Fenofibrate Additive Effects on Lipids (RAFAEL)
Acronym: RAFAEL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment and increase in deployment overseas limiting follow up
Sponsor: Ahmad Slim (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Ahmad Slim, Director, Cardiovascular Research, Brooke Army Medical Center
Organization: Brooke Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2007.122
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Hypertriglyceridemia in Type 4 Hyperlipidemia; Non Diabetic Subjects With Normoglycemia
Keywords: Type 4 hyperlipidemia; Rosiglitazone; Fenofibrate
MeSH Terms: interventions — Rosiglitazone; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Rosiglitazone + Placebo (Active Comparator): Rosiglitazone 8 mg daily + Placebo (Fenofibrate) 145 mg daily for 12 weeks
  Interventions: Drug: Rosiglitazone; Drug: Placebo (Fenofibrate)
- Fenofibrate + Placebo (Active Comparator): Fenofibrate 145mg daily + Placebo (Rosiglitazone) 8mg daily for 12weeks
  Interventions: Drug: Placebo (Rosiglitazone); Drug: Fenofibrate
- Rosiglitazone +Fenofibrate (Experimental): Rosiglitazone 8mg daily + Fenofibrate 145mg daily for 12 weeks
  Interventions: Drug: Rosiglitazone; Drug: Fenofibrate
- Placebo Therapy Daily (Placebo Comparator): Placebo (Rosiglitazone) 8mg daily + Placebo (Fenofibrate) 145 mg daily for 12 weeks
  Interventions: Drug: Placebo (Rosiglitazone); Drug: Placebo (Fenofibrate)

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone 8mg daily for 12 weeks
  Other Names: Avandia
  Arms: Rosiglitazone + Placebo; Rosiglitazone +Fenofibrate
Drug: Placebo (Rosiglitazone) — Placebo (Rosiglitazone) 8mg daily for 12 weeks
  Arms: Fenofibrate + Placebo; Placebo Therapy Daily
Drug: Placebo (Fenofibrate) — Placebo (Fenofibrate) 145 mg daily for 12 weeks
  Arms: Placebo Therapy Daily; Rosiglitazone + Placebo
Drug: Fenofibrate — Fenofibrate 145 mg daily for 12 weeks
  Other Names: Tricor, Triglide, Fenoglide, Lipofen and Lofibra
  Arms: Fenofibrate + Placebo; Rosiglitazone +Fenofibrate

SUMMARY:
The design of the study will be randomized, double blind trial, which will examine the effects of Rosiglitazone on the fasting triglycerides (TG), high-density lipoprotein (HDL), low-density lipoprotein (LDL), and plasma concentrations of apolipoproteins A-I, A-II, and C-III as compared to Fenofibrate and placebo. This study will also assess the synergistic effect of Rosiglitazone and Fenofibrate on the same parameters. Data from this study will help clarify whether Rosiglitazone favorably impacts plasma lipid and lipoprotein concentrations through improving insulin sensitivity and glycemic control, or by directly influencing the synthesis of the apolipoproteins that are responsible for very-low-density lipoprotein (VLDL) and HDL metabolism.

DETAILED DESCRIPTION:
Treatment of patients with type 2 Diabetes Mellitus (DM) consists of reducing hyperglycemia through diet, exercise, oral drug therapy or insulin (1). The Thiazolidinedione (TZDs), which include Troglitazone (withdrawn by the FDA), Rosiglitazone, and Pioglitazone, correct hyperglycemia by increasing insulin sensitivity in both the liver (2, 3) and skeletal muscles (4,5). Although TZDs improve glycemic control in type 2 diabetic subjects, when these agents are administered to non-diabetic subjects they do not affect fasting plasma glucose levels. Nolan et al. (6) observed no effect on the plasma glucose levels of non-diabetic subjects treated with Troglitazone 200 mg twice daily.

Clinical trials using TZDs in type 2 diabetic subjects have observed that these agents also favorably impact plasma lipid and lipoprotein concentrations. A recent study comparing the efficacy of adding Metformin (850 mg, once or twice daily) or Troglitazone (200 mg, once or twice daily) to Glyburide (10 mg, twice daily) on glycemic control in type 2 diabetic patients (n=22), reported that after 4 months of treatment, Metformin did not induce significant changes in LDL-C, LDL size, HDL-C, Triglycerides or Plasminogen Activator Inhibitor-1 (PAI-1), but decreased C-reactive protein (CRP) by 33%. Interestingly, Troglitazone increased the size of LDL and the mean LDL-C level (+10%), but decreased the Triglyceride (-22%) and CRP (-60%) concentrations (7). Following eight weeks of treatment with Rosiglitazone (4mg, twice daily) in 243 type 2 diabetic patients, the mean HDL-C increased by 6% and TG by 2%. The increase in the LDL-C concentration (9%) was accompanied by a shift in small, dense LDL to large, buoyant LDL in 52% of the treated subjects. The shift in LDL size occurred independent of a significant Triglyceride reduction, which is in contrast to several studies reporting that increases in LDL size are significantly correlated with a decrease in the plasma concentrations of total and very low density lipoproteins (VLDL) Triglycerides (8-10).

The mechanism involved in the plasma lipid and lipoprotein changes induced by TZDs remains unclear. It is possible that these agents indirectly alter plasma lipid and lipoprotein levels indirectly by improving insulin sensitivity and glycemic control, or directly by influencing lipoprotein synthesis and/or catabolism.

In type 2 Diabetes Mellitus, hepatic synthesis of Triglycerides is increased and peripheral catabolism is decreased. The primary metabolic defect causing the hypertriglyceridemia is peripheral insensitivity to the action of insulin, accompanied by hyperinsulinemia. The insulin insensitivity inhibits the synthesis and activity of lipoprotein lipase and consequently impairs peripheral catabolism of Triglyceride-rich lipoproteins (VLDL and Chylomicrons) (11-12). Since hepatocytes remain sensitive to the action of insulin, the hyperinsulinemia suppresses beta-oxidation and shunts free fatty acids entering the liver into the synthesis of Triglycerides. Therefore, hepatic production of Triglycerides (i.e. VLDL) is increased at the same time peripheral catabolism is impaired. The result is hypertriglyceridemia with a reciprocal decease in HDL-C concentration. By reducing insulin resistance and plasma insulin levels, TZDs would decrease hepatic Triglyceride production and enhance peripheral catabolism of Triglycerides, resulting in plasma reduction and a reciprocal increase in the HDL-C level.

Recently, it has been recognized that circulating levels of Triglyceride and HDL-C are influenced by the activities of Peroxisome Proliferator Activator Receptors (PPARs). PPARs constitute a super family of nuclear hormone receptors and are ligand-activated transcription factors. When activated, they transmit signals from intra-cellular lipid-soluble factors (e.g. fatty acids, hormones, vitamins) to genes in the nucleus by binding to DNA at specific response elements (13). Three distinct PPARs, termed alpha, beta, and gamma modulate intracellular lipid and glucose metabolism through controlling gene expression when activated (14). Specifically when PPAR-alpha is activated, gene expression for the synthesis of ApoC-III, lipoprotein lipase, ApoA-I and ApoA-II are impacted. ApoC-III is a specific inhibitor of peripheral lipoprotein lipase and competes with ApoE for space on the surface of VLDL. Reduced amounts of ApoC-III will result in a larger representation of ApoE on the VLDL particle, and as a consequence, the ApoE mediated hydrolysis of Triglycerides is enhanced. Activation of PPAR-alpha leads to decrease production of ApoC-III, which in turn results in enhanced clearance of Triglycerides. Activation of PPAR-alpha also increases the synthesis of lipoprotein lipase, which increases Triglyceride catabolism. Gene expression for the synthesis of ApoA-I and ApoA-II is also enhanced by activation of PPAR-alpha, resulting in increase in HDL concentration. Fibric acid derivatives (Gemfibrozil and Fenofibrate) induce their Triglyceride lowering and HDL-C augmenting properties by binding to the PPAR-alpha nuclear receptor.

TZDs are PPAR-gamma ligands that stimulate the gene expression of GLUT1 and GLUT4 (cellular glucose transport proteins) leading to increased insulin sensitivity in the target cells (15,16). The three PPAR receptors possess some degree of structural homology. Therefore, while TZDs have high affinity to PPAR-gamma, they may also bind to a lesser degree to PPAR-alpha or beta. Saliel and Olefsky (17) have determined in cell culture studies that Troglitazone can activate all three PPAR nuclear receptors. Lehmann et al. (18) observed in vitro that TZDs are high affinity ligands for PPAR-gamma yet also bind to PPAR-alpha (to a small degree). Binding PPAR-alpha would directly enhance the catabolism of Triglycerides (i.e. reduced ApoC-III plasma concentrations and increased lipoprotein lipase activity) and increase HDL-C plasma concentration through enhancing the expression of lipoprotein lipase and ApoA-I and ApoA-II. Therefore, administration of TZDs to non-diabetic normoglycemic individuals should not change plasma glucose concentrations, but by binding to PPAR-alpha it would result in decrease in the plasma concentration of ApoC-III, and an increase in ApoA-I and ApoA-II, with a subsequent rise in HDL-C and reduction in Triglyceride concentration.

In a recent animal study assessing Rosiglitazone's mode of action on lipids using male Sprague-Dawley rats, serum total, free and HDL cholesterol concentrations were monitored. In rats given Rosiglitazone, serum Triglyceride levels decreased in a dose-dependent manner, dropping to less than 50% of that of the control rats at the highest dose tested (5 mg/kg/d). Serum glucose concentrations did not change after Rosiglitazone treatment, which is in agreement with previous studies showing that thiazolidinediones do not exert a hypoglycemic action in the normoglycemic, non-diabetic rat. (18)

ELIGIBILITY:
Inclusion criteria:

1. Fasting plasma glucose <100 mg/dl
2. Fasting LDL <160 mg/dl and Triglyceride <400 mg/dl.

Exclusion criteria:

1. Congestive heart failure
2. Evidence of renal impairment (serum creatinine> 1.4mg/dL)
3. Liver disease (ALT and/or AST above the upper level of normal)
4. Known diabetes mellitus or impaired fasting glucose (fasting glucose ≥ 100mg/dL)
5. LDL of ≥160mg/dL and/or triglycerides of ≥400mg/dL
6. Pregnant or breast feeding women
7. Prior history of an acute coronary syndrome, myocardial infarction or revascularization procedures in the past
8. Life-threatening disease with a survival prognosis <3 years
9. Inability to take rosiglitazone and/or fenofibrate
10. Already on statin therapy or have been on statin therapy in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad m slim, MD, Principal Investigator — Brooke Army Medical Center; Laudino Castillo-rojas, MD, Study Chair — Brooke Army Medical Center; Jennifer N Slim, DO, Study Director — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

REFERENCES:
- [Background] O'Rourke CM, Davis JA, Saltiel AR, Cornicelli JA. Metabolic effects of troglitazone in the Goto-Kakizaki rat, a non-obese and normolipidemic rodent model of non-insulin-dependent diabetes mellitus. Metabolism. 1997 Feb;46(2):192-8. doi: 10.1016/s0026-0495(97)90301-2. PMID 9030828
- [Background] Ciaraldi TP, Gilmore A, Olefsky JM, Goldberg M, Heidenreich KA. In vitro studies on the action of CS-045, a new antidiabetic agent. Metabolism. 1990 Oct;39(10):1056-62. doi: 10.1016/0026-0495(90)90166-a. PMID 2120548
- [Background] 5. Troglitazone study group. The metabolic effects of troglitazone in non-insulin dependent diabetes. Diabetes 197; 46:Suppl 1:149A.
- [Background] Nolan JJ, Ludvik B, Beerdsen P, Joyce M, Olefsky J. Improvement in glucose tolerance and insulin resistance in obese subjects treated with troglitazone. N Engl J Med. 1994 Nov 3;331(18):1188-93. doi: 10.1056/NEJM199411033311803. PMID 7935656
- [Background] Chu NV, Kong AP, Kim DD, Armstrong D, Baxi S, Deutsch R, Caulfield M, Mudaliar SR, Reitz R, Henry RR, Reaven PD. Differential effects of metformin and troglitazone on cardiovascular risk factors in patients with type 2 diabetes. Diabetes Care. 2002 Mar;25(3):542-9. doi: 10.2337/diacare.25.3.542. PMID 11874944
- [Background] Coresh J, Kwiterovich PO Jr. Small, dense low-density lipoprotein particles and coronary heart disease risk: A clear association with uncertain implications. JAMA. 1996 Sep 18;276(11):914-5. No abstract available. PMID 8782642
- [Background] Stampfer MJ, Krauss RM, Ma J, Blanche PJ, Holl LG, Sacks FM, Hennekens CH. A prospective study of triglyceride level, low-density lipoprotein particle diameter, and risk of myocardial infarction. JAMA. 1996 Sep 18;276(11):882-8. PMID 8782637
- [Background] Gardner CD, Fortmann SP, Krauss RM. Association of small low-density lipoprotein particles with the incidence of coronary artery disease in men and women. JAMA. 1996 Sep 18;276(11):875-81. PMID 8782636
- [Background] 11. Weinber, R.B. Lipoprotein metabolism: hormone regulation. Hosp. Prac 1987 :June' 15 :125-145.
- [Background] Dunn FL. Hyperlipidemia and diabetes. Med Clin North Am. 1982 Nov;66(6):1347-60. doi: 10.1016/s0025-7125(16)31368-2. No abstract available. PMID 6755099
- [Background] Schoonjans K, Staels B, Auwerx J. Role of the peroxisome proliferator-activated receptor (PPAR) in mediating the effects of fibrates and fatty acids on gene expression. J Lipid Res. 1996 May;37(5):907-25. PMID 8725145
- [Background] Staels B, Dallongeville J, Auwerx J, Schoonjans K, Leitersdorf E, Fruchart JC. Mechanism of action of fibrates on lipid and lipoprotein metabolism. Circulation. 1998 Nov 10;98(19):2088-93. doi: 10.1161/01.cir.98.19.2088. PMID 9808609
- [Background] Bahr M, Spelleken M, Bock M, von Holtey M, Kiehn R, Eckel J. Acute and chronic effects of troglitazone (CS-045) on isolated rat ventricular cardiomyocytes. Diabetologia. 1996 Jul;39(7):766-74. doi: 10.1007/s001250050509. PMID 8817100
- [Background] Ciaraldi TP, Huber-Knudsen K, Hickman M, Olefsky JM. Regulation of glucose transport in cultured muscle cells by novel hypoglycemic agents. Metabolism. 1995 Aug;44(8):976-81. doi: 10.1016/0026-0495(95)90092-6. PMID 7637655
- [Background] Lehmann JM, Moore LB, Smith-Oliver TA, Wilkison WO, Willson TM, Kliewer SA. An antidiabetic thiazolidinedione is a high affinity ligand for peroxisome proliferator-activated receptor gamma (PPAR gamma). J Biol Chem. 1995 Jun 2;270(22):12953-6. doi: 10.1074/jbc.270.22.12953. PMID 7768881
- [Background] Lefebvre AM, Peinado-Onsurbe J, Leitersdorf I, Briggs MR, Paterniti JR, Fruchart JC, Fievet C, Auwerx J, Staels B. Regulation of lipoprotein metabolism by thiazolidinediones occurs through a distinct but complementary mechanism relative to fibrates. Arterioscler Thromb Vasc Biol. 1997 Sep;17(9):1756-64. doi: 10.1161/01.atv.17.9.1756. PMID 9327774
- [Result] 1. American Diabetes association. Standards of medical care for patients with Diabetes Mellitus. Diabetes Care 1997 ;20 : Suppl 1 :55-513.
- [Result] Lee MK, Miles PD, Khoursheed M, Gao KM, Moossa AR, Olefsky JM. Metabolic effects of troglitazone on fructose-induced insulin resistance in the rat. Diabetes. 1994 Dec;43(12):1435-9. doi: 10.2337/diab.43.12.1435. PMID 7958495

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosiglitazone + Fenofibrate: Rosiglitazone 8mg daily + Fenofibrate 145mg daily for 12 weeks
Period: Overall Study
Arm/Group | Rosiglitazone + Placebo | Fenofibrate + Placebo | Rosiglitazone + Fenofibrate | Placebo Therapy Daily
Started | 10 | 10 | 10 | 11
Completed | 8 | 9 | 7 | 10
Not Completed | 2 | 1 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rosiglitazone/Fenofibrate Therapy Daily: Rosiglitazone 8mg once daily and Fenofibrate 145mg once daily for 12 weeks
- Fenofibrate + Placebo: Fenofibrate 145mg once daily for 12 weeks and Placebo (Rosiglitazone 8mg once daily)
- Rosiglitazone + Placebo: Rosiglitazone 8mg once daily and Placebo ( Fenofibrate 145mg once daily)
- Placebo Therapy Daily: Placebo (Rosiglitazone 8mg once daily) and placebo (Fenofibrate 145 mg once daily) for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone/Fenofibrate Therapy Daily | Fenofibrate + Placebo | Rosiglitazone + Placebo | Placebo Therapy Daily | Total
Number analyzed (Participants) | 7 | 9 | 8 | 10 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 7 | 4 | 23
  >=65 years | 1 | 3 | 1 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (9.5) | 61.2 (11.6) | 57.3 (8.4) | 57.4 (11.1) | 56 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 4 | 17
  Male | 3 | 3 | 5 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 8 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Triglyceride (TG) Levels Post Treatment
Description: The reported percent change is the difference between TG levels obtained on initial visit (day 0) and TG levels obtained at final visit (week 12) as per protocol
Time Frame: 12 weeks from initial visit (day 0) to final visit (12 weeks)
Population: Mean percent change post treatment ( unit %). TG was measured using mg/dL units
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Rosiglitazone + Placebo | Fenofibrate + Placebo | Rosiglitazone +Fenofibrate | Placebo Therapy Daily
Number analyzed (Participants) | 8 | 9 | 7 | 10
% change | 7.4 (48.9) | -2.2 (26) | 20 (36.5) | 7.6 (51)

2. Secondary Outcome: Post-treatment Percent Change in High-Density Lipoprotein (HDL) Levels
Description: The reported percent change is the difference between HDL levels obtained on initial visit (day 0) and HDL levels obtained at final visit (week 12) as per protocol
Time Frame: 12 weeks from initial visit (day 0) to final visit (12 weeks)
Measure: Mean (Standard Deviation); unit: % change
Groups:
- Rosiglitazone and Placebo: Rosiglitazone 8 mg daily + Placebo (Fenofibrate) 145 mg daily for 12 weeks
Arm/Group | Rosiglitazone and Placebo | Fenofibrate + Placebo | Rosiglitazone +Fenofibrate | Placebo Therapy Daily
Number analyzed (Participants) | 8 | 9 | 7 | 10
% change | 1.9 (24.6) | 14.5 (21.6) | 5.8 (16.4) | 1.7 (10.5)

3. Secondary Outcome: Post-treatment Percent Change in Low-Density Lipoprotein (LDL) Levels
Description: The reported percent change is the difference between LDL levels obtained on initial visit (day 0) and LDL levels obtained at final visit (week 12) as per protocol
Time Frame: 12 weeks from initial visit (day 0) to final visit (12 weeks)
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Rosiglitazone + Placebo | Fenofibrate + Placebo | Rosiglitazone + Fenofibrate | Placebo Therapy Daily
Number analyzed (Participants) | 8 | 9 | 7 | 10
% change | -0.5 (27.4) | 2.6 (29.3) | 37.3 (141.6) | 13.7 (47.8)

4. Secondary Outcome: Post-treatment Percent Change in Apolipoprotein A-I (Apo AI), Apolipoprotein A-II (Apo AII) and Apolipoprotein C-III (Apo CIII) Levels
Description: Post-treatment median change in Apo AI, Apo AII and Apo CIII levels reported in mg/dL with Interquartile ranges provided
Time Frame: 12 weeks from initial visit (day 0) to final visit (12 weeks)
Measure: Median (Inter-Quartile Range); unit: % Change
Arm/Group | Rosiglitazone + Placebo | Fenofibrate + Placebo | Rosiglitazone +Fenofibrate | Placebo Therapy Daily
Number analyzed (Participants) | 8 | 9 | 7 | 10
% Change
  Apo AI | -1.00 [-34 to 9] | 13 [9 to 18] | 1 [-4 to 12] | 5 [-11 to 16]
  Apo AII | 10.25 [4.90 to 11.50] | 3.4 [2.7 to 7.4] | 7.2 [-2.3 to 8] | -3.5 [-3.6 to 4]
  Apo CIII | 0.30 [0.00 to 1.80] | -4.35 [-7.4 to -2.2] | -5.3 [-6.7 to -3] | -2.3 [-3.7 to 0.7]

5. Secondary Outcome: Mean Levels of Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) at Initial Visit and Final Visit
Description: The mean Levels of AST and ALT measured at initial visit (Day 0) and final visit (Week 12) annotated as AST 1, AST 12, and ALT 1 and ALT 12, respectively.
Time Frame: 12 weeks from initial visit (day 0) to final visit (12 weeks)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rosiglitazone + Placebo | Fenofibrate + Placebo | Rosiglitazone +Fenofibrate | Placebo Therapy Daily
Number analyzed (Participants) | 8 | 9 | 7 | 10
mg/dl
  AST 1 (aspartate aminotransferase [10-35 U/L]) | 24.00 (11.091) | 25.25 (7.517) | 24.30 (5.870) | 19.88 (5.249)
  AST 12 (aspartate aminotransferase [15-37 U/L]) | 30.29 (9.810) | 26.50 (7.964) | 19.70 (2.584) | 17.88 (6.139)
  ALT 1 (alanine aminotransferase [6-60 U/L]) | 28.14 (13.957) | 25.88 (15.394) | 24.10 (10.429) | 20.88 (6.643)
  ALT 12 (alanine aminotransferase [6-60 U/L]) | 27.43 (10.358) | 26.38 (11.916) | 21.10 (8.647) | 14.88 (3.523)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: These are the adverse events reported during the monitoring period in 41 initial participants contributing to partially to drop out of 7 participants and the final data reported in the results section of only 34 participants.
Groups:
- Rosiglitazone/Fenofibrate Therapy Daily: Rosiglitazone 8mg po daily + Fenofibrate 145 mg po daily for 12 weeks
  These are the adverse events reported in population who continued the 12 weeks of therapy as well as the population that dropped out.
- Rosiglitazone + Placebo: Rosiglitazone 8mg po daily + Placebo (Fenofibrate 145 mg po daily) for 12 weeks
  These are the adverse events reported in population who continued the 12 weeks of therapy as well as the population that dropped out.
- Fenofibrate + Placebo: Fenofibrate 145 mg po daily for 12 weeks= Placebo (Rosiglitazone 8mg po daily)
  These are the adverse events reported in population who continued the 12 weeks of therapy as well as the population that dropped out.
- Placebo Therapy Daily: Rosiglitazone (placebo) once daily and Fenofibrate (placebo)once daily for 12 weeks
  These are the adverse events reported in population who continued the 12 weeks of therapy as well as the population that dropped out.
Arm/Group | Rosiglitazone/Fenofibrate Therapy Daily | Rosiglitazone + Placebo | Fenofibrate + Placebo | Placebo Therapy Daily
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/10 | 1/10 | 0/11
Other Adverse Events (participants affected / at risk) | 8/10 | 4/10 | 2/10 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone/Fenofibrate Therapy Daily (N=10) | Rosiglitazone + Placebo (N=10) | Fenofibrate + Placebo (N=10) | Placebo Therapy Daily (N=11)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone/Fenofibrate Therapy Daily (N=10) | Rosiglitazone + Placebo (N=10) | Fenofibrate + Placebo (N=10) | Placebo Therapy Daily (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aching legs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stiff Neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Severe Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Severe sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tiredness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pressure behind left eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen Ankles (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
First, the study was terminated early per FDA recommendations restricting rosiglitazone use. Second, recruitment of patients was slow due to deployment restraints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less